CLINICAL TRIAL: NCT06474143
Title: Evaluation of the Clinical Performance of Apneal®, a Medical Device on Smartphone, for Sleep Apnea-hypopnea Syndrome Diagnosis studY
Brief Title: Evaluation of the Clinical Performance of Apneal®, a Medical Device on Smartphone, for Sleep Apnea-hypopnea Syndrome Diagnosis.
Acronym: EASY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C23-80; 2023-A02144-41 (Registry Identifier: IDRCB)
Record Dates: First submitted 2024-02-07; First posted 2024-06-25 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Sleep Apnea Syndromes
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Each patient will wear the device and polysomnograph at the same time
Masking Description: Polysomnography results not available to device
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epxerimental (Experimental): Patients will wear the device during their polysomnographic recording
  Interventions: Device: Apneal device

INTERVENTIONS:
Device: Apneal device — Patients will wear a smartphone with the Apneal Application on their chest, while they perform polysomnography

SUMMARY:
The goal of this clinical trial is to test the ability of the Apneal application in diagnosing sleep apnea in adult patients.

Participants will be asked to wear the Apneal device during their fulll-night sleep test (polysomnography, the gold standard for sleep apnea)

ELIGIBILITY:
Inclusion Criteria:

* Individuals, men or women, aged over 18 and with no upper age limit;
* Individuals for whom PSG is indicated as part of routine care, regardless of indication.
* Individuals willing and able to comply with study requirements;
* Individuals with a declared total sleep time of at least 6 hours, as recommended by AASM for PSG analysis.
* Individuals affiliated to social security or beneficiary of such a scheme if applicable according to the local regulation ;
* Voluntary individuals who have provided oral and written consent after being informed by the research investigator.

Exclusion Criteria:

* Individuals with active implantable medical devices (e.g. electronic heart implant, electrical neurophysiological stimulator…);
* Individuals with mechanical heart valves;
* Individuals with chest deformity preventing the phone to be correctly placed on the chest
* Individuals with uncontrolled psychiatric conditions impairing their ability to fully consent to the study
* Individuals suffering from epilepsy or an associated disorder;
* Individuals suffering from a moderate to severe valvular disease;
* Individuals under CPAP treatment during the participation.
* Individuals suffering from a nervous system disorder that causes unintended or uncontrollable movements, other than periodic leg movement syndrome and restless leg syndrome.
* Refusal to participate in the study at any time during the clinical investigation;
* Individuals in period of exclusion from another protocol or currently participating in another interventional research study;
* Individuals not able to understand and speak the official language of the research center;
* Vulnerable individuals according to local legislation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Performance of Apneal® in categorizing SAHS severity using AHI | through study completion, an average of 1 year
  The primary endpoint of this study is the performance of Apneal® in categorizing SAHS severity in four classes compared to PSG: normal (AHI < 5), mild (5 ≤ AHI < 15), moderate (15 ≤ AHI < 30), and severe (AHI ≥ 30)

SECONDARY OUTCOMES:
Correlation between AHI from Apneal and AHI from PSG | through study completion, an average of 1 year
  The endpoint requires to assess the performances of Apneal® against PSG first. The ground truth and predicted severities will be established and compared for each included individual.
Correlation between AHI from Apneal and AHI from nocturnal polygraphy | through study completion, an average of 1 year
  The endpoint requires to assess the performances of Apneal® against polygraphy channels derived from PSG first. The ground truth and predicted severities will be established and compared for each included individual.
Correlation between AHI from apneal and ODI from nocturnal oximetry | through study completion, an average of 1 year
  The endpoint requires to assess the performances of Apneal®, against nocturnal oximetry, . The ground truth and predicted severities will be established and compared for each included individual.
  The comparison of Apneal® performance with nocturnal oximetry for sleep apnea screening will be conducted using ROC analysis.
Correlation between AHI from Apneal and NoSAS score | through study completion, an average of 1 year
  The endpoint requires to assess the performances of Apneal® in screening OSAS, against NoSAS . The ground truth and predicted severities will be established and compared for each included individual. The first step is to output a score for each of these methods :
  * AHI for Apneal®
  * NoSAS score
  The comparison of Apneal® with NoSAS for sleep apnea screening will be conducted using ROC analysis.
Correlation between AHI from Apneal and STOPBANG score | through study completion, an average of 1 year
  The endpoint requires to assess the performances of Apneal® in screening OSAS, against NoSAS . The ground truth and predicted severities will be established and compared for each included individual. The first step is to output a score for each of these methods :
  * AHI for Apneal®
  * STOPBANG score
  The comparison of Apneal® with STOPBANG for sleep apnea screening will be conducted using ROC analysis.
Correlation between AHI from Apneal and Berlin score | through study completion, an average of 1 year
  The endpoint requires to assess the performances of Apneal® in screening OSAS, against Berlin questionnaire. The ground truth and predicted severities will be established and compared for each included individual. The first step is to output a score for each of these methods :
  * AHI for Apneal®
  * Berlin score
  The comparison of Apneal® with Berlin for sleep apnea screening will be conducted using ROC analysis.
Correlation between AHI from Apneal and Epworth sleepiness scale (ESS) score | through study completion, an average of 1 year
  The endpoint requires to assess the performances of Apneal® in screening OSAS, against Berlin questionnaire. The ground truth and predicted severities will be established and compared for each included individual. The first step is to output a score for each of these methods :
  * AHI for Apneal®
  * Epworth sleepiness scale (ESS) score
  The comparison of Apneal® with ESS for sleep apnea screening will be conducted using ROC analysis.
The classification of sleep epochs into three categories : wake, REM sleep and NREM sleep (N1, N2 or N3). | through study completion, an average of 1 year
  The ground truth (from PSG) and predicted (from Apneal®) sleep stages classification will be established and compared for each included individual after :
  * the PSG and Apneal® data are recorded during the inclusion visit (sleep study)
  * the PSG sleep stages are estimated by the scorer in the centralized center, following AASM guidelines
  * the ground truth sleep stages are output from these estimations or the adjudication committee if there is a disagreement between the two first scorers.
  * Apneal® sleep stages are predicted automatically by the Apneal® algorithm. Sleep stages from Apneal® and PSG are compared using accuracy of the binary classifications.
The segmentation of the night in snores and non-snores periods | through study completion, an average of 1 year
  Segmentations of Apneal® and manual scoring of the recorded sound, by a sleep technologist in the centralized scoring center, will be compared.
Heart rate | through study completion, an average of 1 year
  The heart rate predicted by Apneal®, compared with the heart rate derived from ECG on PSG.
Autonomic sleep fragmentation | through study completion, an average of 1 year
  The autonomic sleep fragmentation index, which is the average amount of autonomic arousals per hour of sleep. It will be estimated by Apneal® and compared with the autonomic sleep fragmentation index derived from ECG on PSG.
Central apnea index | through study completion, an average of 1 year
  amount of central apneas per hour of sleep. Apneal® will estimate this index, and it will be compared with the central apnea index measured on PSG.
Position detection | through study completion, an average of 1 year
  The segmentation of the participant's position in 6 categories: supine, left, right, prone, sitting and standing. Segmentation of Apneal® and PSG will be compared. position on PSG will be manually scored, position on Apneal is predicted automatically by the Apneal® algorithm.
Wake/night detection | through study completion, an average of 1 year
  The segmentation of the night as wake and sleep predicted by Apneal® and manually scored on PSG will be compared.
Medicoeconomic study | through study completion, an average of 1 year
  The estimated relative difference between the costs of visits, with and without Apneal® in the clinical pathway
Medicoeconomic study | through study completion, an average of 1 year
  The estimated relative difference between the number of visits, with and without Apneal® in the clinical pathway

CONTACTS AND LOCATIONS:
Locations (1):
- Centre du sommeil, hôpital Bichat, Paris, France